CLINICAL TRIAL: NCT02691741
Title: Clinical Investigation of Visual Function After Bilateral Implantation of Two Presbyopia-Correcting Trifocal IOLs
Brief Title: Clinical Investigation of Visual Function After Bilateral Implantation of Two Presbyopia-Correcting Trifocal Intraocular Lenses (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILH297-P003
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TFNT00 (Experimental): AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL, bilateral implantation
  Interventions: Device: AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL
- 839MP (Active Comparator): AT LISA® tri IOL, bilateral implantation
  Interventions: Device: AT LISA® tri IOL

INTERVENTIONS:
Device: AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL — Trifocal IOL(near, intermediate, distance) implanted for long-term use over the lifetime of the cataract patient
  Other Names: Model TFNT00
  Arms: TFNT00
Device: AT LISA® tri IOL — Trifocal IOL(near, intermediate, distance) implanted for long-term use over the lifetime of the cataract patient
  Other Names: Model 839MP
  Arms: 839MP

SUMMARY:
The purpose of this study is to clinically evaluate the visual performance of two commercially available presbyopia-correcting Trifocal IOLs.

DETAILED DESCRIPTION:
Subjects will attend a total of 9 visits (6 postoperative) over a 7 month period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral cataracts with planned clear cornea cataract removal;
* Able to comprehend and willing to sign informed consent and complete all required postoperative follow-up procedures;
* Calculated lens power between 13.0 and 30.0 Diopters (D);
* Preoperative Best-corrected distance visual acuity (BCDVA) worse than 0.20 logMAR (ie, 0.22 logMAR or worse) in at least one eye;
* Potential postoperative BCDVA of 0.20 logMAR or better in both eyes. Note: Subjects with any pathology that could reduce visual potential should not be enrolled in this trial;
* Preoperative regular corneal astigmatism of < 1.00 D, in both eyes;
* Clear intraocular media other than cataract in both eyes;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Reasonably expected to require an ocular surgical treatment at any time during the study (other than YAG capsulotomy);
* Previous refractive surgery or planned refractive surgery procedures throughout the entire duration of participation in the clinical study (including, but not limited to LASIK, astigmatic keratotomy and limbal relaxing incisions);
* Clinically significant corneal abnormalities including corneal dystrophy, inflammation or edema;
* Amblyopia;
* Previous corneal transplant;
* Any recurrent severe anterior or posterior segment inflammation of any etiology, and/or history of any disease producing an intraocular inflammatory reaction;
* Rubella, congenital, traumatic, or complicated cataracts;
* Glaucoma (uncontrolled or controlled with medication);
* Degenerative eye disorders;
* History of or current retinal conditions or predisposition to retinal conditions, previous history of, or a predisposition to, retinal detachment or presence of diabetic retinopathy;
* Optic nerve atrophy;
* Expected to require retinal laser treatment;
* Color vision deficiencies;
* Pregnant or lactating (current or planned during the course of the study);
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA, Study Director — Alcon, a Novartis Company

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 15 study centers located in Australia (3), Brazil (3), Spain (3), Denmark (2), Colombia (2), United Kingdom (1), and the Netherlands (1).
Pre-assignment Details: Of the 215 enrolled, 26 subjects were exited as screen failures and 1 subject died prior to randomization. This reporting group includes all randomized subjects (188).
Period: Overall Study
Arm/Group | TFNT00 | 839MP
Started (Randomized subjects) | 94 | 94
All-Implanted Analysis Set (All subjects with successful test or control article bilateral implantation) | 93 | 89
Best-Case Analysis Set (All subjects successfully implanted, at least 1 post-op visit, no mac. degen., no major deviations) | 86 | 85
Safety Analysis Set (All subjects with attempted implantation (successful or aborted after contact with the eye)) | 93 | 89
Completed | 93 | 87
Not Completed | 1 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: All-Implanted Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | TFNT00 | 839MP | Total
Number analyzed (Participants) | 93 | 89 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (9.29) | 65.6 (9.56) | 65.9 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 55 | 112
  Male | 36 | 34 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White or Caucasian | 42 | 39 | 81
  Race/Ethnicity: Black or African American | 2 | 2 | 4
  Race/Ethnicity: Asian | 3 | 8 | 11
  Race/Ethnicity: American Indian or Native American | 0 | 0 | 0
  Race/Ethnicity: Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Race/Ethnicity: Multi-Racial | 0 | 2 | 2
  Race/Ethnicity: Other | 44 | 38 | 82

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Binocular Uncorrected Intermediate Visual Acuity (UCIVA) (60cm) at Day 120-180
Description: VA was tested binocularly (both eyes together) with no refractive correction in place using an early treatment diabetic retinopathy study (ETDRS) chart set at 60 cm. VA was measured in "logarithm of the minimum angle of resolution" (logMAR), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Day 120-180 from second eye implantation
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 93 | 89
logMAR | 0.053 (0.0134) | 0.115 (0.0139)
Statistical Analysis 1: Comparison: TFNT00 vs 839MP; Test type: Non-Inferiority — Non-inferiority is demonstrated if the upper confidence limit of the two-sided 90% confidence interval on the treatment difference is less than 0.1 logMAR unit; Mean Difference (Final Values) = -0.061, 90% CI 2-sided [-0.093 to -0.029], Standard Error of Mean 0.0193

2. Secondary Outcome: Least Squares Mean Binocular UCIVA (60cm) at Day 120-180
Description: VA was tested binocularly with no refractive correction in place using an ETDRS chart set at 60 cm. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Day 120-180 from second eye implantation
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 93 | 89
logMAR | 0.053 (0.0134) | 0.115 (0.0139)
Statistical Analysis 1: Comparison: TFNT00 vs 839MP; Test type: Superiority; p = 0.002, Repeated Measures Analysis of Variance; Mean Difference (Final Values) = -0.061, 90% CI 2-sided [-0.093 to -0.029], Standard Error of Mean 0.0193

3. Secondary Outcome: Least Squares Mean Binocular Uncorrected Distance VA (4m) at Day 120-180
Description: VA was tested binocularly with no refractive correction in place using an ETDRS chart set at 4 meters. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Day 120-180 from second eye implantation
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 93 | 89
logMAR | 0.015 (0.0109) | 0.004 (0.0113)
Statistical Analysis 1: Comparison: TFNT00 vs 839MP; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.019 to 0.043], Standard Error of Mean 0.0157
Statistical Analysis 2: Comparison: TFNT00 vs 839MP; Test type: Superiority; p = 0.455, Repeated Measures Analysis of Variance

4. Secondary Outcome: Least Squares Mean Binocular Uncorrected Near VA (40cm) at Day 120-180
Description: VA was tested binocularly with no refractive correction in place using an ETDRS chart set at 40 cm. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity.
Time Frame: Day 120-180 from second eye implantation
Population: All-Implanted Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 93 | 89
logMAR | 0.083 (0.0116) | 0.133 (0.0121)
Statistical Analysis 1: Comparison: TFNT00 vs 839MP; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.051, 90% CI 2-sided [-0.078 to -0.023], Standard Error of Mean 0.0168
Statistical Analysis 2: Comparison: TFNT00 vs 839MP; Test type: Superiority; p = 0.003, Repeated Measures Analysis of Variance

5. Secondary Outcome: Mean Photopic Binocular Defocus Curve at Day 120-180
Description: A defocus curve is created by multiple measurements of one's visual acuity (VA) at different spherical powers. VA was measured in logMAR. A lower logMAR value indicates better visual acuity. No statistical test was performed.
Time Frame: Day 120-180 from second eye implantation
Population: This analysis population includes all subjects with eyes successfully implanted with the test or control article that had at least one postoperative visit, and with no macular degeneration at any time, and no major protocol deviations (Best-Case Analysis Set), with data available.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 86 | 81
logMAR
  0.0 Diopter (D) | -0.048 (0.0811) | -0.069 (0.0831)
  -0.5D | 0.016 (0.0835) | -0.018 (0.0951)
  -1.0D | 0.093 (0.0993) | 0.048 (0.1207)
  -1.5D | 0.038 (0.0983) | 0.084 (0.1111)
  -2.0D | 0.011 (0.0859) | 0.117 (0.1039)
  -2.5D | 0.027 (0.1013) | 0.063 (0.1399)
  -3.0D | 0.118 (0.1297) | 0.077 (0.1241)
  -3.5D | 0.231 (0.1252) | 0.206 (0.1415)
  -4.0D | 0.338 (0.1319) | 0.364 (0.1302)
  -4.5D | 0.469 (0.1417) | 0.532 (0.1240)
  -5.0D | 0.586 (0.1292) | 0.644 (0.1048)

6. Secondary Outcome: Mean Photopic Without Glare Binocular Distance Contrast Sensitivity at Day 120-180
Description: Contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly in lighted conditions with distance manifest correction in place and uncorrected, with no glare source illumination. Contrast sensitivity was assessed at spatial frequencies of 3, 6, 12, and 18 cycles per degree (CPD) and reported in log units. A higher numeric value represents better contrast sensitivity. No statistical test was performed.
Time Frame: Day 120-180 from second eye implantation
Population: Best-Case Analysis Set, with available data
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 86 | 81
log units
  3 CPD | 1.720 (0.2025) | 1.735 (0.1894)
  6 CPD | 1.860 (0.2635) | 1.831 (0.2699)
  12 CPD | 1.482 (0.3853) | 1.496 (0.4328)
  18 CPD | 1.021 (0.3778) | 1.022 (0.4197)

7. Secondary Outcome: Mean Photopic With Glare Binocular Distance Contrast Sensitivity at Day 120-180
Description: Contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly in lighted conditions with distance manifest correction in place and uncorrected, with glare source illumination. Contrast sensitivity was assessed at spatial frequencies of 3, 6, 12, and 18 CPDs and reported in log units. A higher numeric value represents better contrast sensitivity. No statistical test was performed.
Time Frame: Day 120-180 from second eye implantation
Population: Best-Case Analysis Set, with data available
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 86 | 81
log units
  3 CPD | 1.721 (0.2041) | 1.754 (0.2225)
  6 CPD | 1.790 (0.3282) | 1.797 (0.3538)
  12 CPD | 1.434 (0.4616) | 1.426 (0.4570)
  18 CPD | 1.007 (0.3769) | 1.033 (0.4316)

8. Secondary Outcome: Mean Mesopic Without Glare Binocular Distance Contrast Sensitivity at Day 120-180
Description: Contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly in dim to dark conditions with distance manifest correction in place and uncorrected, with no glare source illumination. Contrast sensitivity was assessed at spatial frequencies of 1.5, 3, 6, and 12 CPDs and reported in log units. A higher numeric value represents better contrast sensitivity. No statistical test was performed.
Time Frame: Day 120-180 from second eye implantation
Population: Best-Case Analysis Set with data available
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 86 | 81
log units
  1.5 CPD | 1.611 (0.2293) | 1.600 (0.2226)
  3 CPD | 1.648 (0.3115) | 1.682 (0.2639)
  6 CPD | 1.667 (0.4284) | 1.676 (0.4243)
  12 CPD | 1.208 (0.5262) | 1.227 (0.5307)

9. Secondary Outcome: Mean Mesopic With Glare Binocular Distance Contrast Sensitivity at Day 120-180
Description: Contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly with distance manifest correction in place and uncorrected, with glare source illumination. Contrast sensitivity was assessed at spatial frequencies of 1.5, 3, 6, and 12 CPDs and reported in log units. A higher numeric value represents better contrast sensitivity. No statistical test was performed.
Time Frame: Day 120-180 from second eye implantation
Population: Best-Case Analysis Set, with data available
Measure: Mean (Standard Deviation); unit: log units
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 86 | 81
log units
  1.5 CPD | 1.579 (0.2581) | 1.538 (0.2568)
  3 CPD | 1.642 (0.2696) | 1.682 (0.2642)
  6 CPD | 1.550 (0.4791) | 1.607 (0.4898)
  12 CPD | 1.146 (0.5623) | 1.175 (0.6062)

10. Secondary Outcome: Subject Satisfaction Recorded at Day 120-180
Description: At the Month 6 Visit, subjects responded to the question: "Given your current postoperative vision, if you had to do it all over would you have the same lens implanted again?". Responses were reported as a percentage of subjects. No statistical test was performed.
Time Frame: Day 120-180 from second eye implantation
Population: All-Implanted Analysis Set with data available
Measure: Number; unit: percentage of subjects
Arm/Group | TFNT00 | 839MP
Number analyzed (Participants) | 93 | 87
percentage of subjects
  Yes | 95.7 | 96.6
  No | 3.2 | 2.3
  Missing | 1.1 | 1.1

ADVERSE EVENTS:
Time Frame: IOL implantation through study completion, an average of 7 months
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device. AEs were obtained through solicited comments from subjects by the Investigators. Safety Analysis Set. "At risk" population for ocular AEs is reported in units of eyes.
Groups:
- TFNT00 - 1st Eye: First eye implanted with AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL
- TFNT00 - 2nd Eye: Second eye implanted with AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL
- TFNT00 - Systemic: Subjects implanted with AcrySof® IQ PanOptix™ Presbyopia-Correcting IOL in at least one eye
- 839MP - 1st Eye: First eye implanted with AT LISA® tri IOL
- 839MP - 2nd Eye: Second eye implanted with AT LISA® tri IOL
- 839MP - Non-Study Eye: Eyes not meeting study inclusion/exclusion criteria
- 839MP - Systemic: Subjects implanted with AT LISA® tri IOL in at least one eye
Arm/Group | TFNT00 - 1st Eye | TFNT00 - 2nd Eye | TFNT00 - Systemic | 839MP - 1st Eye | 839MP - 2nd Eye | 839MP - Non-Study Eye | 839MP - Systemic
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/93 | 0/93 | 0/89 | 0/87 | 0/2 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/93 | 2/93 | 3/89 | 2/87 | 0/2 | 0/89
Other Adverse Events (participants affected / at risk) | 8/93 | 8/93 | 0/93 | 7/89 | 3/87 | 0/2 | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TFNT00 - 1st Eye (N=93) | TFNT00 - 2nd Eye (N=93) | TFNT00 - Systemic (N=93) | 839MP - 1st Eye (N=89) | 839MP - 2nd Eye (N=87) | 839MP - Non-Study Eye (N=2) | 839MP - Systemic (N=89)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intra-ocular injection (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Intraocular lens implant (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TFNT00 - 1st Eye (N=93) | TFNT00 - 2nd Eye (N=93) | TFNT00 - Systemic (N=93) | 839MP - 1st Eye (N=89) | 839MP - 2nd Eye (N=87) | 839MP - Non-Study Eye (N=2) | 839MP - Systemic (N=89)
Halo vision (Eye disorders) | 5 | 5 | 0 | 2 | 2 | 0 | 0
Posterior capsule opacification (Eye disorders) | 3 | 3 | 0 | 5 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT02691741/SAP_000.pdf
  • Study Protocol (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02691741/Prot_001.pdf